CLINICAL TRIAL: NCT05262582
Title: Randomized Open Label Two Arms Cohort Study to Evaluate Curative Effect and Quality of Life of Single Port and Two Ports Robotic Assisted Thoracic Surgery for Thymectomy
Brief Title: Comparison of Single Port and Two Ports Robotic Assisted Thoracic Surgery for Thymectomy
Acronym: RATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Lei Jiang, principal investigator, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jianglei4
Record Dates: First submitted 2022-01-16; First posted 2022-03-02 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Thymoma; Myasthenia Gravis Associated With Thymoma; Thymectomy
Keywords: Thymoma; Myasthenia Gravis; Thymectomy; Robotic Assisted Thoracic Surgery
MeSH Terms: conditions — Thymoma; Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymectomy performed with sigle port RATS (Experimental): The incision is performed in the 5-6th intercostal space under the breast folds without violating the mammalian tissue. This port is used for the camera and both arms simultaneously.
  Interventions: Procedure: Sigle port RATS
- Thymectomy performed with two ports RATS (Active Comparator): The incision is performed in the 4th intercostal space along anterior axillary fossa, for the camera and left arm. The other incision is subxiphoid longitudinal incision about 4cm for the right arm.
  Interventions: Procedure: Two ports RATS

INTERVENTIONS:
Procedure: Sigle port RATS — The incision is performed in the 5-6th intercostal space under the breast folds without violating the mammalian tissue. This port is used for the camera and both arms simultaneously.
  Arms: Thymectomy performed with sigle port RATS
Procedure: Two ports RATS — The incision is performed in the 4th intercostal space along anterior axillary fossa, for the camera and left arm. The other incision is subxiphoid longitudinal incision about 4cm for the right arm.
  Arms: Thymectomy performed with two ports RATS

SUMMARY:
Recently, robotic-assisted thoracic surgery (RATS) has become into as an alternative approach to either, open surgery or video-assisted thoracoscopic surgery. The superiorities of RATS have been reported in series studies, such as intuitive movements, tremor filtration, more degrees of manipulative freedom, motion scaling, and high-definition stereoscopic vision.

However, the currently reported robotic thymectomy used 3 ports. Theoretically, less incisions may bring faster postoperative recovery, lighter postoperative pain and higher postoperative quality of life. The investigators have successfully performed robotic thymectomy through 2 ports and even 1 port. However, the potential benefit of less ports robotic thymectomy has not been verified through well-designed cohort study, so this clinical trial has been designed.

DETAILED DESCRIPTION:
The gold standard technique for thymectomy used to be transsternal approach. Advancements in modern technology bring many evolutions in minimally invasive surgery such as Video-assisted thoracic surgery (VATS) thymectomy gained popularity after 2000s. Recently, robotic-assisted thoracic surgery (RATS) has become into as an alternative approach to either, open surgery or video-assisted thoracoscopic surgery. The superiorities of RATS have been reported in series studies, such as intuitive movements, tremor filtration, more degrees of manipulative freedom, motion scaling, and high-definition stereoscopic vision.

However, the currently reported robotic thymectomy used 3 ports. Theoretically, less incisions may bring faster postoperative recovery, lighter postoperative pain and higher postoperative quality of life. The investigators have successfully performed robotic thymectomy through 2 ports and even 1 port. However, the potential benefit of less ports robotic thymectomy has not been verified through well-designed cohort study, so this clinical trial has been designed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Myasthenia Gravis and(or) thymoma need to perform thymectomy.
2. Agree to accept Robotic Assisted Thoracic Surgery and have signed informed consent.

Exclusion Criteria:

1. Cardiopulmonary function cannot tolerate thoracoscopic surgery or exist other contraindication.
2. Thymic carcinoma.
3. Thoracic deformity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Post operation pain | 1 month after surgery
  Measured with Visual Analogue Score (VAS-score)，the minimum value is 1, the maximum value is 10, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Surgical bleeding | During operation
  Surgical bleeding measured with milliliter
Operation duration | During operation
  Operation duration measured with minute
Quality of life after surgery | 6 months
  Measured with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core30 (EORTC QLQ-C30 questionnaire), the higher scores mean a better outcome.
Curative effect | 5 years
  Disease free survival 5 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng M, Wang X, Chen C, Tan S, Liu W, Yu F. Report on 153 sequential three-incision robotic-assisted pulmonary resections by a single surgeon: technical details and learning curve. J Thorac Dis. 2020 Mar;12(3):741-748. doi: 10.21037/jtd.2019.12.116. PMID 32274140
- [Background] Kaba E, Cosgun T, Ayalp K, Alomari MR, Toker A. Robotic thymectomy-a new approach for thymus. J Vis Surg. 2017 May 8;3:67. doi: 10.21037/jovs.2017.03.28. eCollection 2017. PMID 29078630
- [Background] Curcio C, Scaramuzzi R, Amore D. Robotic-assisted thoracoscopic surgery thymectomy. J Vis Surg. 2017 Nov 7;3:162. doi: 10.21037/jovs.2017.10.01. eCollection 2017. PMID 29302438
- [Background] Luzzi L, Corzani R, Ghisalberti M, Meniconi F, De Leonibus L, Molinaro F, Paladini P. Robotic surgery vs. open surgery for thymectomy, a retrospective case-match study. J Robot Surg. 2021 Jun;15(3):375-379. doi: 10.1007/s11701-020-01109-z. Epub 2020 Jul 6. PMID 32632562